CLINICAL TRIAL: NCT07242196
Title: Comparison of the Analgesic Effects of Ultrasound-Guided Transversalis Fascia Plane Block and Transversus Abdominis Plane Block in Pediatric Laparoscopic Surgery
Brief Title: Transversalis Fascia Plane Versus Transversus Abdominis Plane Block for Postoperative Analgesia in Children
Status: Recruiting | Type: Observational
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Burçin Alaçam, MD, Anesthesiology Specialist, Sakarya University
Other Study IDs: E-43012747-050.04-513206-484
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Analgesia; Transversus Abdominis Plane (TAP) Block; Transversalis Fascia Plane Block; Pediatric Surgical Procedures; Laparoscopic Abdominal Surgeries
Keywords: transversus abdominis plane block; transversalis fascia plane block; pediatrics; laparoscopic abdominal surgery; postoperative analgesia
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Transversalis Fascia Plane Block: Patients in this group will receive an ultrasound-guided transversalis fascia plane block prior to surgery. The local anesthetic will be injected between the transversus abdominis muscle and the deep transversalis fascia at the level of the posterior axillary line, targeting the proximal portions of the T12 and L1 nerves. This technique aims to provide effective analgesia for the anterolateral abdominal wall and to extend sensory blockade coverage compared to traditional Transversus Abdominis Plane block. Postoperative pain, additional analgesic requirements, and duration of analgesia will be monitored and recorded.
  Interventions: Other: Postoperative analgesia
- Group Transversus Abdominis Plane Block: Patients in this group will receive an ultrasound-guided transversus abdominis plane (TAP) block prior to surgery. The local anesthetic will be administered between the internal oblique and transversus abdominis muscles, typically providing analgesia in the T10-L1 dermatomes. This group will serve as a comparative control to assess the relative efficacy of the TAP block versus the transversalis fascia plane block in managing postoperative pain. Postoperative Visual Analog Scale scores, need for rescue analgesics, and duration of analgesia will be recorded.
  Interventions: Other: Postoperative analgesia

INTERVENTIONS:
Other: Postoperative analgesia — Postoperative analgesia will be assessed using the Visual Analog Scale (VAS) at predefined time points following surgery: 1, 2, 4, 8, 12, and 24 hours postoperatively. Pain evaluation will be performed both at rest and during movement (e.g., coughing or mobilization).
  Additional analgesics will be administered according to a standardized protocol: intravenous paracetamol (15 mg/kg/dose, every 6 hours as needed) will be given if VAS ≥ 4. Rescue analgesia requirements, including timing and dosage, will be recorded for each patient.
  The primary aim of this assessment is to compare the analgesic efficacy of ultrasound-guided transversalis fascia plane block and transversus abdominis plane block in pediatric patients undergoing laparoscopic surgery. Duration of analgesia, postoperative VAS scores, and need for rescue analgesics will be documented to determine the relative effectiveness of each block technique.

SUMMARY:
This prospective clinical study aims to compare the postoperative analgesic efficacy of the ultrasound-guided transversalis fascia plane block (TFPB) and the transversus abdominis plane (TAP) block in pediatric patients undergoing laparoscopic surgery. Effective and long-lasting postoperative analgesia is essential for patient and parental satisfaction in pediatric anesthesia. With recent advances in ultrasound technology, regional anesthesia techniques have become increasingly utilized in pediatric practice.

In the TAP block, local anesthetic is injected between the internal oblique and transversus abdominis muscles, providing analgesia typically between Torachal vertebra 10 (T10) and Lumbar vertebra (L1) dermatomes. The transversalis fascia plane block, developed as a modification of this approach, targets the proximal portions of the T12 and L1 nerves by depositing local anesthetic between the transversus abdominis muscle and the transversalis fascia, potentially offering wider sensory coverage.

This study compares both blocks in terms of postoperative pain scores, duration of analgesia, and requirement for rescue analgesics in children undergoing laparoscopic surgery. The results are expected to contribute to the optimization of regional anesthesia techniques and improve pain management strategies in pediatric surgical patients.

DETAILED DESCRIPTION:
In pediatric anesthesia, achieving effective and long-lasting analgesia is essential for ensuring the satisfaction of both pediatric patients and their parents. To guarantee this, many pediatric anesthesiologists have incorporated various regional anesthesia techniques into their daily clinical practice. Advances in technology have enabled the use of many regional anesthesia techniques across diverse clinical settings.

The transversus abdominis plane (TAP) block is an interfascial plane block technique in which a local anesthetic is typically administered, under ultrasound guidance, between the internal oblique and transversus abdominis muscles. Although several approaches have been described for this block, all involve the injection of anesthetic into this interfascial layer, providing analgesia from the T10 to L1 dermatomes. With the widespread adoption of ultrasound technology in pediatric practice, this technique and related fascial plane blocks have become increasingly popular.

The transversalis fascia plane (TFP) block was developed as a technique aiming to block more thoracic nerves. In this approach, local anesthetic is injected between the transversus abdominis muscle and the deep transversalis fascia at the level of the posterior axillary line, targeting the proximal portions of the T12 and L1 nerves. The blockade extends medially toward the inner surface of the quadratus lumborum muscle, thereby providing a more effective block of the anterolateral abdominal wall.

The aim of this study is to compare the postoperative analgesic efficacy of ultrasound-guided transversalis fascia plane block and transversus abdominis plane block in pediatric patients undergoing laparoscopic surgery. The primary outcome of the study is the evaluation of postoperative pain using validated pediatric pain assessment scales at defined postoperative intervals. The secondary outcomes include the assessment of additional analgesic requirements, the duration of postoperative analgesia provided by each block, and any block-related complications. Furthermore, this research aims to enhance knowledge regarding regional anesthesia applications in pediatric patients and provide scientific contributions to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 6 months to 16 years
* Classified as ASA physical status I or II
* Scheduled to undergo laparoscopic surgery under general anesthesia

Exclusion Criteria:

* Patients classified as ASA physical status III or IV
* Known allergy or hypersensitivity to local anesthetic agents
* Presence of bleeding diathesis or coagulation disorders
* Infection at the injection site or local skin lesions preventing block application

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population will include pediatric patients aged 6 months to 16 years who are scheduled to undergo elective laparoscopic surgery under general anesthesia. All participants will be classified as ASA physical status I or II according to the American Society of Anesthesiologists classification. Patients with ASA III-IV status, known allergy to local anesthetic agents, bleeding diathesis or coagulation disorders, and infection at the injection site will be excluded. Eligible patients of both sexes will be enrolled, and healthy volunteers will not be included. Participants will be randomly assigned to receive either an ultrasound-guided transversalis fascia plane block or a transversus abdominis plane block for postoperative analgesia. The study aims to represent the typical pediatric population undergoing minimally invasive abdominal surgery under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Assessment (Visuel Analog Scale) | At 1, 2, 4, 8, 12, and 24 hours after surgery.
  The primary outcome is the comparison of the analgesic efficacy of the transversalis fascia plane block and the transversus abdominis plane block in pediatric laparoscopic surgery, measured using the Visuel Analog Scale (VAS). The Visual Analog Scale is a standardized tool used to quantify the intensity of pain. It consists of a 10-centimeter horizontal line representing a continuous range of pain levels. The minimum score is 0, indicating no pain, and the maximum score is 10, indicating the worst imaginable pain. Higher scores reflect worse outcomes, meaning greater pain intensity. Participants are asked to mark a point on the line that best represents the severity of their pain, and the distance from the zero point is measured in centimeters to obtain the final score.

SECONDARY OUTCOMES:
Duration of Analgesia | 24 hours after surgery
  Time from block administration to the first report of pain Visuel Analog Scale (VAS ≥ 4) or request for rescue analgesia.
Rescue Analgesic Requirement | 24 hours after surgery
  The number and total dose of additional analgesic medications (Intravenosus paracetamol 15 mg/kg as needed for Visual Analog Scale (VAS) ≥ 4) administered within 24 hours postoperatively.
Incidence of Block-Related Complications | 24 hours after surgery
  Any block-related adverse events (e.g., hematoma, infection, local anesthetic toxicity) observed perioperatively or postoperatively.
Patient and Parental Satisfaction | 24 hours after surgery
  Satisfaction with postoperative pain control, assessed using a 5-point Likert scale at 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University-Anesthesiology and Reanimation Department, Sakarya, Serdivan, Turkey (Türkiye)

REFERENCES:
- [Result] Fredrickson MJ, Paine C, Hamill J. Improved analgesia with the ilioinguinal block compared to the transversus abdominis plane block after pediatric inguinal surgery: a prospective randomized trial. Paediatr Anaesth. 2010 Nov;20(11):1022-7. doi: 10.1111/j.1460-9592.2010.03432.x. PMID 20964768